CLINICAL TRIAL: NCT02960087
Title: A Randomized Phase II Trial Evaluating High Dose Rate Brachytherapy and Low Dose Rate Brachytherapy as Monotherapy in Localized Prostate Cancer
Brief Title: Phase II High Dose Brachytherapy and Low Dose Rate Brachytherapy as Monotherapy in Localized Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR19
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 LDR (Active Comparator): Low Dose Rate (LDR) brachytherapy with I-125 to a total dose of 144 Gy
  Interventions: Radiation: Low dose rate brachytherapy
- Arm 3 HDR (Active Comparator): High Dose Rate brachytherapy: 27 Gy in 2 fractions
  Interventions: Radiation: High dose rate brachytherapy

INTERVENTIONS:
Radiation: Low dose rate brachytherapy — I-125 to a total dose of 144 Gy
  Arms: Arm 1 LDR
Radiation: High dose rate brachytherapy — 27 Gy in 2 fractions
  Arms: Arm 3 HDR

SUMMARY:
The purpose of this study is to evaluate the dose of High Dose Rate (HDR) brachytherapy chosen for this study as well as a commonly used alternate form of brachytherapy called low dose rate (or seed) brachytherapy. Investigators would like to understand how these treatments control the prostate cancer and look at their short and long term treatment related side effects.

The dose of radiation for HDR brachytherapy for this study has been changed since the study started. Other studies using the dose of radiation for HDR brachytherapy that was originally chosen for this study (Arm 2) found that this dose of radiation may be linked to a greater chance of the cancer coming back in the prostate. Therefore since March 2020, for new participants entering the study, a new HDR brachytherapy arm with a higher amount of radiation given over two doses will be tested in this study

DETAILED DESCRIPTION:
Radiation therapy is an accepted treatment to help manage low and intermediate risk prostate cancer. Radiation therapy can be given using machines that are outside the body (called "image guided external beam radiation therapy") or by brachytherapy, which is a form of radiation therapy where the radiation source is placed directly into the prostate gland near the tumour. The standard or usual treatments for low or intermediate risk prostate cancer are low dose-rate (LDR) brachytherapy which involves placing radioactive seeds in the prostate which deliver radiation over several months, image guided external beam radiation therapy (IGRT), or IGRT plus high dose-rate (HDR) brachytherapy boost.

High Dose-Rate (HDR) brachytherapy is another type of brachytherapy which delivers a high dose of radiation to the tumour over a period of minutes. The radiation is delivered under computer control through flexible needles, which are temporarily inserted into the prostate. This form of radiotherapy targets cancer cells within the prostate gland. HDR brachytherapy is another type of radiotherapy for prostate cancer that has the potential to help target your cancer more accurately while causing fewer side effects compared with standard radiation therapy. HDR brachytherapy is an option for treatment in some hospitals now but the best dose of radiation is still unknown. This study is testing a new dose of radiation for HDR brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate diagnosed within the last 9 months. Patients on active surveillance with evidence of disease progression are eligible to the protocol as long as they meet the eligibility criteria and have a recent prostate biopsy (within 9 months).
* Patients with localized prostate cancer are eligible according to the following guidelines:

  • TNM classification:
  * Clinical stage T1-T2 and Gleason 6 and PSA <20 ng/mL
  * Clinical stage T1-T2 and Gleason 7 (3+4) and PSA < 15 ng/mL and ≤ 50% of positive nontargeted cores in patients who undergo systematic biopsy
* Eastern Cooperative Oncology Group status 0-1.
* Bone scan and pelvic CT scan/MRI within the last 6 months at the discretion of the treating physician.
* Patient must be ≥ 18 years of age.
* Judged to be medically fit for brachytherapy.
* Prostate volume by Trans-rectal Ultrasound (TRUS) or Magnetic Resonance Imaging (MRI) ≤ 60 cc within the last 6 months.
* American Urological Association (AUA) score ≤ 20 (alpha blockers allowed) within the last 4 weeks.
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in either English or French.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrolment in the trial to document their willingness to participate.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre.
* In accordance with CCTG policy, protocol treatment is to begin within 12 weeks of patient randomization.
* Patients must be willing to take precautions to prevent pregnancy while on study.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

* Prior or current bleeding diathesis.
* Previous androgen deprivation therapy (ADT).
* Alpha-reductase inhibitors (ARIs) within 90 days of randomization.
* Radical surgery for carcinoma of the prostate, prior pelvic radiation, prior chemotherapy for prostate cancer, prior TURP, prior cryosurgery of the prostate.
* Evidence of metastatic disease (radiology investigations at the discretion of the treating physician).
* Any serious active or co-morbid medical conditions, laboratory abnormality, psychiatric illness, active or uncontrolled infections, or serious illnesses or medical conditions that would prevent the patient from participating or to be managed according to the protocol (according to investigator's decision).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of HDR and LDR brachytherapy on prostate cancer control as defined by 48 month PSA values | 48 months
  The primary endpoint of the study is prostate cancer control rate at 48 months. It is defined as the PSA <0.4ng/ml at 48 months. One sample binomial test will be used to test the 48 months disease control rate for each arm

SECONDARY OUTCOMES:
Disease-free survival | 7 years
Number and severity of adverse events | 7 years
  Acute and long term toxicity and safety including lower urinary tract symptoms
Quality of Life of patient and partner utilizing EPIC, PROMIS and R-DAS fatigue short form | 7 years
Economic Analysis | 7 years
  Resource utilization and economic indices of treatment administration

OTHER OUTCOMES:
Establish a comprehensive tumour bank linked to a clinical database for further studies of predictive and prognostic biomarkers in prostate cancer | 7 years
PSA Progression - PSA nadir +2 ng/ml will be used to define biochemical failure and can only be declared at 36 months or beyond due to the phenomenon of PSA bounce | 7 years
PSA nadir - Date PSA nadir +2 ng/ml is reached | 7 years
Local disease progression - Clinically suspicious change in DRE with biopsy confirmation of progression or Urethral obstruction or bleeding necessitating a trans-urethral resection (TURP) only if resected tissue demonstrates malignancy | 7 years
Regional disease progression - Prostate cancer progression involving the lymph nodes below the bifurcation of the common iliac arteries. | 7 years
Distant disease progression - Evidence of prostate cancer by radiology or cytology or histology at sites remote from the prostate | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Morton, Study Chair — Sunnybrook Health Sciences, Toronto ON; Eric Vigneault, Study Chair — Hotel Dieu de Quebec, Montreal, QC
Locations (7):
- Canada (7):
  - London Health Sciences Centre Research Inc., London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No